CLINICAL TRIAL: NCT03585829
Title: Comparison of the Risk of Complications and the Quality of Life During Ramadan Fasting in Patients With Corticotrope Deficiency Treated Either by Hydrocortisone or by Prednisolone
Brief Title: Ramadan Fasting in Patients With Corticotrope Deficiency Treated Either by Hydrocortisone or by Prednisolone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Melika Chihaoui, Principal investigator, University Tunis El Manar
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 100
Record Dates: First submitted 2018-05-16; First posted 2018-07-13 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Corticotropin Deficiency; Fasting
Keywords: treatment; quality of life; hypoglycemia
MeSH Terms: conditions — Adrenocorticotropic hormone deficiency; Fasting; Hypoglycemia | interventions — Hydrocortisone; Prednisolone

STUDY DESIGN:
Intervention Model Description: crossover clinical trial
Who Masked: Participant, Care Provider
Masking Description: the treatment has been put in capsules with the same size and color
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrocortisone (Active Comparator): hydrocortisone 20 mg per day: 15 mg at pre-dawn meal and 5 mg at dinner
  Interventions: Drug: Hydrocortisone
- prednisolone (Active Comparator): Prednisolone 5 mg at pre-dawn meal and a placebo (starch) at dinner
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Hydrocortisone — at a substitutive dosage
  Other Names: Cortef*
  Arms: hydrocortisone
Drug: Prednisolone — at a substitutive dosage
  Other Names: Vitapred*
  Arms: prednisolone

SUMMARY:
Selected patients will be randomised to either hydrocortisone or prednisolone. Each treatment period is of 14 days. Abnormal clinical symptoms, blood glucose and quality of life will be monitored.

DETAILED DESCRIPTION:
* Selection of the patients who meet the inclusion and non inclusion criteria.
* Detailed explanations about the study to the patients.
* Signature of the informed consent by the patients.
* Randomisation of the patients by drawing lots into two groups; group AB who will receive treatment A during 14 days (period 1) then treatment B during 14 days (period 2) and group BA who will receive treatment B during 14 days (period 1) then treatment A during 14 days (period 2).
* Each patient will receive a daily follow-up sheet, a quality of life questionnaire, a glucometer with test strips and the treatment in different bottles for each period of the study.
* The daily follow-up sheet concerns habits during Ramadan (eating, sleeping), the occurrence of complications and blood glucose monitoring. Daily blood glucose monitoring is requested at midday, before dinner and if a malaise occurs. A detailed questionnaire on abnormal symptoms that might occur during fasting have to be fulfilled for each malaise.
* Quality of life will be evaluated using AddiQol questionnaire translated in Tunisian dialect. Patients have to complete the questionnaire before the fasting month and at the end of each period of treatment.
* Treatment is presented in the form of capsules with the same colour and size. Patients have to take one capsule at dinner and one capsule at pre-dawn meal. Patients will receive either hydrocortisone 15mg at pre-dawn meal and 5mg at dinner (sunset) (treatment A) or prednisolone 5mg at pre-dawn meal and a placebo (starch) at dinner (treatment B).
* During the study, patients will be in regular phone contact with a responsible of the study for any information or problem.
* At the end of the study, the completed follow-up sheets and questionnaires will be picked up.

ELIGIBILITY:
Inclusion Criteria:

* Known corticotrope deficiency treated by 20mg hydrocortisone per day.
* Age: 18-70 years
* patients who are willing to fast Ramadan 2018 and who voluntary accept to participate in the study.

Non inclusion criteria:

Patients with either diabetes mellitus, hypertension, diabetes insipidus, severe organ damage (renal, cardiac, pulmonary, hepatic), neoplasia, psychiatric disease, epilepsy or pregnant or breast-feeding women.

Exclusion Criteria:

The occurrence of any of the non inclusion criteria during the study. The occurrence of a severe malaise.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Occurence of complications | during the fourteen days treatment period
  fatigue, asthenia, symptoms of hypoglycemia, symptoms of dehydration, hypoglycemia on blood glucose monitoring

SECONDARY OUTCOMES:
score of quality of life | during the fourteen days treatment period
  using a questionnaire (AddiQol)

CONTACTS AND LOCATIONS:
Overall Officials: Hedia Slimane, MD, Study Chair — University Tunis El Manar
Locations (1):
- University Tunis El Manar, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No